CLINICAL TRIAL: NCT00991250
Title: A Multi-centre, Two-arm, Randomized, Open, Phase II Study Investigating SentoClone® Compared to Reference Treatment in Advanced Malignant Melanoma
Brief Title: SentoClone® Compared to Reference Treatment in Advanced Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SentoClone AB (Industry)
Responsible Party: Freddi Lewin, Medical director, SentoClone AB
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mel-Swe-01 2009-12-17; EudraCT No: 2008-007515-33
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SentoClone® (Experimental): SentoClone®: Specific tumour-reactive lymphocytes located in lymph nodes directly draining primary tumours or metastases are identified and expanded. These lymphocytes are infused to the patient to treat metastatic disease.
  Interventions: Biological: SentoClone®
- Temodal® or Dacarbazine Medac® (Active Comparator): To be decided by each centre as one of the following:
  1. Temodal® (temozolomide)
  2. Dacarbazine Medac® (dacarbazine) The reference treatment regimen should follow the general guiding principles for each of the two reference treatments.
  Interventions: Drug: Temodal® or Dacarbazine Medac®

INTERVENTIONS:
Biological: SentoClone® — SentoClone® are autologous tumour-reactive lymphocytes which are expanded and infused to the patient, where they have the opportunity to seek out and attack the primary tumour and metastases. The first step is to identify the tumour draining lymph node(s), which is done in parallel to surgical resection of the primary tumour or metastasis. The sentinel and/or metinel node(s), the initial meeting place between tumour antigen and the immune system, are further dissected and collected during the surgery. The lymphocytes are extracted from the collected lymph nodes and expanded in vitro, the lymphocytes are thereafter stimulated with tumour extract and returned to the patient intravenously as an autologous cell transfusion. The administered volume will be 100 ml for cell densities less than 3x106 cells/ml and 200 ml for cell densities of 3x106 cells/ml or more.
  Arms: SentoClone®
Drug: Temodal® or Dacarbazine Medac® — Dacarbazine (5-[3,3-Dimethyl-1-triazenyl]imidazole-4-carboxamide) is a widely used systemic treatment against advanced malignant melanoma. Dacarbazine is a cytostatic agent, which inhibits tumour growth by interfering with DNA-synthesises. The DNA-synthesis is inhibited by alkylation of the DNA molecule; however, it is unclear whether dacarbazine has other cytostatic impacts on cell mechanisms. Dacarbazine is inactive until liver passage, the liver converts dacarbazine to its reactive metabolites MTIC and HMMTIC, which alkylate DNA. Dacarbazine is light sensitive and needs to be administered intravenously.
  A newer analogue to dacarbazine, temozolomide (Temodal®), has been developed for oral administration. Temodal® is administered in capsules and is rapidly absorbed reaching peak concentrations after 20 minutes. Temodal® is converted to MTIC at physiological pH, the same reactive molecule as dacarbazine is metabolized to in the liver.
  Other Names: DTIC; Dacarbazine; Temozolomide
  Arms: Temodal® or Dacarbazine Medac®

SUMMARY:
The purpose of this study is to elucidate whether SentoClone® gives improved treatment responses in patients with advanced malignant melanoma in comparison to established reference treatment(s).

DETAILED DESCRIPTION:
Malignant melanoma is one of the most common cancer forms worldwide and WHO estimates 132,000 new cases each year. The incidence rate vary up to 150-fold between different regions and ethnicities, the highest rates are found in emigrated Caucasian populations (e.g. Australia and New Zealand).

There are few therapy alternatives for advanced malignant melanomas. At present, dacarbazine (Dacarbazine Medac®) is the most commonly used therapy. Immunotherapy with IL-2 and IFN is an alternative, but it is associated with multiple side effects. Hence, there remains a considerable need for alternative treatments.

By using SentoClone®, autologous tumour-reactive lymphocytes are expanded and infused to the patient, where they have the opportunity to seek out and attack the primary tumour and metastases. The first step is to identify the tumour draining lymph node(s), which is done in parallel to surgical resection of the primary tumour or metastasis. The sentinel and/or metinel node(s), the initial meeting place between tumour antigen and the immune system, are further dissected and collected during the surgery.

In this study SentoClone® will be compared with Dacarbazine Medac® and Temodal® which are currently regarded as standard first-line therapies in advanced malignant melanoma.

ELIGIBILITY:
Inclusion Criteria

To be eligible for inclusion in this study, the patients must fulfil all of the following criteria:

1. Surgically incurable stage III or IV malignant melanoma
2. At least one measurable lesion
3. WHO performance status 0-1
4. Life expectancy > 3 months
5. Diagnosed metastasis
6. One tumour draining lymph node surgically accessible
7. Measurable tumour manifestation after the harvest of tumour tissue and sentinel/metinel nodes(1)
8. Signed informed consent

(1) Should be fulfilled after surgery (visit 2) for patients randomised to SentoClone®.

Exclusion Criteria

To be eligible for inclusion in this study the patients must not meet any of the following criteria:

1. Known allergy against used trace substance patent blue and/or albumin technetium (Nanocoll) 2. Known allergy against gentamicin and/or phenol red 3. Any condition (medical, social, psychological or legal) that influences adequate information negatively or is considered to be a problem for the patient to cope with treatment and follow-up 4. Aplastic anaemia or myelofibrosis 5. Previous treatment with temozolomide or dacarbazine, or any other chemotherapy during the last 3 months 6. Disease progression following treatment with temozolomide or dacarbazine more than 3 months back(1) 7. Previous radiotherapy of target lesion(s) or tumour draining lymph nodes which will be used for lymphocyte extraction(2) 8. Ongoing systemic steroid treatment or other treatment influencing immune defence 9. History of other malignant tumour disease apart from adequately treated basalioma or squamous cell carcinoma of the skin more than 5 years ago 10. Positive test(s) for HIV and/or Hepatitis B and/or Hepatitis C and/or syphilis 11. Condition or disease which could influence the result of the study or which indicates that the patient runs risks by participating in this study 12. Participation in any other clinical study, involving other investigational methods or products that may influence the results of this trial, within 30 days prior to participating in this trial

1. Patients who responded on the treatment, terminated the treatment at least 3 months prior to the study, and later progressed do not fulfill exclusion criterion 6
2. Irradiated lesions are not considered to be measurable and are therefore not suitable as target lesions. Lesions which have been irradiated but shown progression are considered as measurable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Tumour response rate, defined as complete response (CR) or partial response (PR) (i.e. at least partial response) measured using the RECIST (Response Evaluation Criteria in Solid Tumours) criteria. | At baseline and 18, 26 and 34 weeks after treatment

SECONDARY OUTCOMES:
Progression-free survival | From baseline to week 34 after initiated treatment
Overall survival | From baseline to week 34 after initiated treatment
Time to tumour progression | From baseline to week 34 after initiated treatment
Disease-free survival | From baseline to week 34 after initiated treatment
Time to treatment failure | From baseline to week 34 after initiated treatment
Duration of response | From baseline to week 34 after initiated treatment
Correlation between tumour response and tumour marker S100 | From baseline to week 34 after initiated treatment
Proportion of patients showing toxic symptoms according to CTCAE criteria | From baseline to week 34 after initiated treatment
Quality of life (EQ-5D and QLQ-C30) | From baseline to week 34 after initiated treatment
Adverse Events (AEs) classified according to seriousness, causality, and intensity, clinically significant deviations in vital signs, clinical chemistry, and haematology | From baseline to week 34 after initiated treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ingvar, MD, Principal Investigator — Lund University Hospital
Locations (5):
- Sweden (5):
  - Lunds Universitetssjukhus, Lund, Skåne County
  - Södersjukhuset, Stockholm, Stockholm County
  - Karolinska Sjukhuset, Stockholm, Stockholm County
  - Norrlands Universitetssjukhus, Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County